CLINICAL TRIAL: NCT05365256
Title: Impact of Virtual Reality on the Mental Health of Patients Undergoing Adjuvant Treatment for Colorectal Cancer VIRECAPS2
Brief Title: Impact of Virtual Reality on the Mental Health of Patients Undergoing Adjuvant Treatment for Colorectal Cancer
Acronym: VIRECAPS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A02382-39
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Cancer of Colon; Virtual Reality
Keywords: virtual reality; Colorectal cancer; Quality of life; Mental Health
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard time occupation of treatment period (Active Comparator): habitual distraction of patients during chemotherapy sessions authorized as part of routine care (doing nothing, discussion, reading, games, etc.).
  Interventions: Behavioral: Standard distraction during chemotherapy treatment period
- time occupation of treatment period by virtual reality (Experimental): Use of virtual reality as a distraction during chemotherapy sessions. A virtual reality headset will be worn for 15 minutes per hour of treatment (with a maximum of three sessions per cycle of chemotherapy)
  Interventions: Behavioral: Virtual distraction during chemotherapy treatment period

INTERVENTIONS:
Behavioral: Standard distraction during chemotherapy treatment period — habitual distraction of patients during chemotherapy sessions authorized as part of routine care
  Arms: Standard time occupation of treatment period
Behavioral: Virtual distraction during chemotherapy treatment period — A virtual reality headset will be worn for 15 minutes per hour of treatment
  Arms: time occupation of treatment period by virtual reality

SUMMARY:
The increase in the survival of cancer patients and the incidence of cancers leads to a rapid increase in the number of people living after a diagnosis of cancer.

Occupation during chemotherapy treatment time has been identified as an excellent way to support cancer patients. Studies show that distraction interventions increase tolerance to treatment, by decreasing the importance given to negative stimuli associated with chemotherapy and increasing pleasurable emotions.

In this context, virtual reality (VR) is a promising intervention for patients receiving chemotherapy. VR is considered a powerful painkiller, even more effective than other distractors, such as movies or video games for example.

Several studies have shown short-term beneficial effects of integrating VR in patients undergoing chemotherapy. This intervention would help patients better adhere to and tolerate treatment. Considering that positive emotions could be one of the underlying processes necessary for the effectiveness of VR, it would be possible to support the cancer patient towards better overall well-being thanks to these new technologies.

Investigators can therefore ask themselves the question of the impact that VR used during chemotherapy can have on the adaptation of patients to the disease and its treatments as well as on their psychological distress in the medium and long term.

DETAILED DESCRIPTION:
The increase in the survival of cancer patients and the incidence of cancers leads to a rapid increase in the number of people living after a diagnosis of cancer. Supporting people during and after treatment is an element of the third Cancer Plan (2014-2019) promoting the emergence of innovations for the benefit of patients as well as the implementation of global and personalized actions of support, and wishing to reduce the impact of cancer on personal life.

Occupation during chemotherapy treatment time has been identified as an excellent way to support cancer patients. Studies show that distraction interventions (progressive relaxation, guided imagery, cognitive distractions such as reading, humor, listening to music, watching a movie, etc.) increase tolerance to treatment, by decreasing the importance given to negative stimuli associated with chemotherapy and increasing pleasurable emotions.

In this context, virtual reality (VR) is a promising intervention for patients receiving chemotherapy. It makes it possible to modulate the attentional and emotional processes responsible for physiological and psychic reactions (pain, psychological distress, anxiety). VR is considered a powerful painkiller, even more effective than other distractors, such as movies or video games for example.

Several studies have shown short-term beneficial effects of integrating VR in patients undergoing chemotherapy. This intervention would help patients better adhere to and tolerate treatment. Considering that positive emotions could be one of the underlying processes necessary for the effectiveness of VR, it would be possible to support the cancer patient towards better overall well-being thanks to these new technologies.

Investigators can therefore ask themselves the question of the impact that VR used during chemotherapy can have on the adaptation of patients to the disease and its treatments as well as on their psychological distress in the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years of age.
* Patient with colorectal cancer treated with adjuvant chemotherapy.
* Chemotherapy naïve patient
* Patient speaking and understanding French and able to complete the questionnaires.
* Affiliated patient or beneficiary of a social security scheme.
* Patient having been informed of the research and having signed a free and informed consent

Exclusion Criteria:

* Patient participating in another clinical study
* Patient with a history or progressive psychiatric illness
* Patient with severe visual and hearing impairment
* Patient not supporting the wearing of the virtual reality headset
* Patient who is unable to undergo medical monitoring for geographical, social or psychological reasons
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Level of psychological well-being | 6 months
  Total score from WEMWBS scale

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lantheaume, Dr, Principal Investigator — Ramsay Santé - Hôpital Privé Drôme
Locations (1):
- Hôpital Privé Drôme Ardèche, Guilherand-Granges, AURA, France

REFERENCES:
- [Result] Banos RM, Espinoza M, Garcia-Palacios A, Cervera JM, Esquerdo G, Barrajon E, Botella C. A positive psychological intervention using virtual reality for patients with advanced cancer in a hospital setting: a pilot study to assess feasibility. Support Care Cancer. 2013 Jan;21(1):263-70. doi: 10.1007/s00520-012-1520-x. Epub 2012 Jun 13. PMID 22688373
- [Result] Chirico A, Lucidi F, De Laurentiis M, Milanese C, Napoli A, Giordano A. Virtual Reality in Health System: Beyond Entertainment. A Mini-Review on the Efficacy of VR During Cancer Treatment. J Cell Physiol. 2016 Feb;231(2):275-87. doi: 10.1002/jcp.25117. PMID 26238976
- [Result] Cohn MA, Fredrickson BL, Brown SL, Mikels JA, Conway AM. Happiness unpacked: positive emotions increase life satisfaction by building resilience. Emotion. 2009 Jun;9(3):361-8. doi: 10.1037/a0015952. PMID 19485613
- [Result] Bani Mohammad E, Ahmad M. Virtual reality as a distraction technique for pain and anxiety among patients with breast cancer: A randomized control trial. Palliat Support Care. 2019 Feb;17(1):29-34. doi: 10.1017/S1478951518000639. Epub 2018 Sep 10. PMID 30198451
- [Result] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Result] Schneider SM, Kisby CK, Flint EP. Effect of virtual reality on time perception in patients receiving chemotherapy. Support Care Cancer. 2011 Apr;19(4):555-64. doi: 10.1007/s00520-010-0852-7. Epub 2010 Mar 26. PMID 20336327
- [Result] Schneider SM, Hood LE. Virtual reality: a distraction intervention for chemotherapy. Oncol Nurs Forum. 2007 Jan;34(1):39-46. doi: 10.1188/07.ONF.39-46. PMID 17562631
- [Result] Tugade MM, Fredrickson BL, Barrett LF. Psychological resilience and positive emotional granularity: examining the benefits of positive emotions on coping and health. J Pers. 2004 Dec;72(6):1161-90. doi: 10.1111/j.1467-6494.2004.00294.x. PMID 15509280